CLINICAL TRIAL: NCT01215019
Title: 20% Mannitol vs 3% Hypertonic Saline in the Treatment of Intracranial Hypertension in Patients With Traumatic Brain Injury: A Double-blinded, Randomized Trial
Brief Title: Osmotic Therapy for Treatment of Intracranial Hypertension for Traumatic Brain Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding; not subjects enrolled
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1004-10
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Mannitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): 20% Mannitol
  Interventions: Drug: Mannitol
- Arm 2 (Active Comparator): 3% sodium chloride
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Mannitol — 20% Mannitol, 1-5 doses as needed to control ICP
  Arms: Arm 1
Drug: NaCl — 3% sodium chloride injection, 1-5 doses, as needed to control ICP
  Other Names: 3% sodium chloride injection
  Arms: Arm 2

SUMMARY:
Osmotic therapy is a mainstay in the treatment of intracranial hypertension after traumatic brain injury.This study proposes to compare two hypertonic saline agents in patients with traumatic brain injury.

DETAILED DESCRIPTION:
Osmotic therapy is a mainstay in the treatment of intracranial hypertension after traumatic brain injury. Despite sparse concrete evidence of beneficial effects on patient outcome, it has been widely accepted by treating physicians that osmotic therapy is effective, at least in helping control elevated intracranial pressure (ICP), and control of ICP has been shown to improve outcome. Mannitol is the most commonly utilized agent. It is widely available, effective, and has a low side-effect profile. Large doses for long term periods have been shown to be safe, but its usefulness is limited by elevation of serum osmolarity and potential alteration in renal function, and its efficacy seems to diminish with repeated doses. Rebound intracranial hypertension has been reported after discontinuation of large doses. Other hypertonic agents such as urea and glycerol are no longer used.

More recently, hypertonic saline (HTS) solutions of various concentrations have become available, and have been shown in several animal research studies and small human trials to be safe and effective in the management of intracranial hypertension. HTS does not cross the blood-brain barrier, and has the ability to improve intravascular volume without the osmotic diuresis effect of mannitol. Several institutions routinely use HTS solutions in the management of traumatic brain injuries, and the use of both mannitol and HTS is common. Additionally longer-term use of HTS is not as restricted by plasma osmolarity. There have been several small trials comparing the two agents, but these studies have been relatively poorly controlled and therefore reached limited conclusions. At our institution both agents (in the forms of 20% mannitol and 3% sodium chloride) are used routinely, with no particular rationale for one over the other. There is suggestion that one agent may be better than the other, but this has not been explicitly tested in humans.

It is our hypothesis that HTS and mannitol both adequately treat intracranial hypertension, but that HTS may have additional benefits of allowing more frequent and/or longer-term dosing, and volume expansion without osmotic diuresis (thereby improving the patient's overall fluid state, potentially decreasing morbidity).

We propose a study of patients with acute traumatic brain injury requiring osmotic therapy to control elevated ICP, comparing the use of 20% mannitol to 3% sodium chloride (NaCl).

Specific Aims:

Primary Goal:

Assess efficacy of 20% mannitol versus 3% NaCl in controlling elevated ICP in acute traumatic brain injury

Secondary Goals:

Assess effects on hemodynamic parameters (mean arterial pressure, cerebral perfusion pressure, central venous pressure and volume status) Assess effects on serum sodium and osmolarity Assess effects on patient outcomes at discharge

ELIGIBILITY:
Inclusion Criteria:

* All hemodynamically stable patients aged 18-65 presenting with acute traumatic brain injury requiring monitoring of intracranial pressure (ICP) will be screened for randomization.

Exclusion Criteria:

* Patients with known pre-existing renal abnormalities or serum creatinine greater than or equal to 2.0mg/dl will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Assess efficacy of 20% mannitol versus 3% MaCl in controlling elevated intracranial pressure in acute traumatic brain injury | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. Rodgers, MD, Principal Investigator — Indiana University
Locations (1):
- Wishard Memorial Hospital, Indianapolis, Indiana, United States